CLINICAL TRIAL: NCT03625336
Title: MR Imaging of Prostatic Calcifications
Status: Withdrawn | Type: Observational
Why Stopped: study on hold for an undetermined time
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Janesh Lakhoo, Radiology Resident, Vanderbilt University Medical Center
Other Study IDs: VR52257
Record Dates: First submitted 2018-08-07; First posted 2018-08-10 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Prostate Calcification
Keywords: prostate; calcification; MRI
MeSH Terms: conditions — Calcinosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prostate Calcifications: Men with prostate calcifications
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — An MRI will be obtained utilizing 3 different MRI sequences

SUMMARY:
Prostate calcifications can limit evaluation of the prostate due to artifact on MRI, and can limit therapy by blocking therapeutic ultrasound. There is definite need to develop and validate MR imaging techniques to visualize focal calcifications, especially for focal therapy planning and monitoring. It will obviate need for CT correlation, help in focal ablation modality selection and give true relative location of the calcification vis-à-vis visualized tumor without need for fusion. Imaging calcifications and evaluation of their effect on high energy ultrasound will help us define clinically significant calcifications. It is also the first step in development of techniques to mitigate effect of calcifications on therapeutic ultrasound. Multiple promising MR sequences are available for possible evaluation of the prostate and this study looks to evaluate the ability of those MRI sequences at detecting and accurately quantifying prostatic calcifications compared to CT, the current gold standard.

DETAILED DESCRIPTION:
The traditional prostate cancer (PCa) screening, diagnosis, and treatment options comprising of prostate-specific antigen (PSA) testing, random transrectal ultrasound (TRUS) biopsy, and prostatectomy/radiation have significant limitations. PSA is a nonspecific test, which is elevated in many benign situations. The American Cancer Society's estimate of 161,360 new cases of PCa in the United States in 2017 is a significantly lower number than that of 2016 (180,890) and 2015 (220,800), mostly due to the United States Preventative Services Taskforce (USPTF) recommendations against routine PSA testing. Random TRUS biopsy is notorious for the conundrum of overdiagnosis of low-risk PCa and under detection of high-risk PCa. Random biopsy of the prostate to diagnose or exclude cancer is performed nearly 1,000,000 times annually in the United States, most frequently as a result of elevated PSA. Less than one-third of these are positive. Both prostatectomy and radiation are associated with high risks of incontinence and impotence. Many patients with low- and intermediate-risk disease unnecessarily undergo these aggressive treatment options.

There is considerable ongoing effort to improve the deficiencies in the diagnostic and treatment approaches. For example, better screening methodologies are being developed, including strategies on how to incorporate prostate magnetic resonance imaging (MRI) into the screening algorithm. The improvement in prostate MRI techniques and advent of targeted biopsy techniques has enabled physicians to actually see and target the risk driving "index" lesion. In the treatment realm, a wide range of minimally invasive modalities has been tested for whole-gland, partial-gland, and focal treatments. Therapeutic ultrasound is a popular FDA-approved, nonsurgical, "no-needle" ablative therapy that does not use ionizing radiation. Theoretically, therapeutic ultrasound has the potential to markedly reduce treatment-related complications that affect urinary and sexual function. While prostate therapeutic ultrasound is FDA-approved, it is not reimbursed by major insurance carriers and its efficacy is still under investigation.

As with diagnostic ultrasound, therapeutic ultrasound can be blocked by calcifications leading to sub-optimal delivery of the thermal dose to the tumor foci. Also, if MR guidance is being used, the most commonly used method of MR thermometry (proton resonance frequency shift) doesn't work well in areas with calcifications. Currently, most major manufacturers of prostate therapeutic ultrasound equipment have limitations related to calcifications:

1. Sonablate (transrectal ultrasound guided high-intensity focused ultrasound (HIFU) device, FDA approved) user manual states that "As with any ultrasound technology, significant changes in tissue density such as calcifications and/or cysts (depending on size) may have an effect on ultrasound attenuation and overall energy and may impact the patient's suitability for treatment".
2. Ablatherm (FDA approved, similar to Sonablate): While calcifications in ablation volume are not a contra-indication for prostate ablation with this device, it can treat only small prostates with larger prostates (> 24 mm AP) requiring cytoreduction via transurethral resection (TURP) presumably removing most calcifications which are usually found along the pseudocapsule.
3. TULSA-PRO: This is a transurethral MR guided device which is currently undergoing clinical trials. Calcifications greater than 1 cm are a contra-indication for whole gland ablation. However, even smaller calcifications can prevent heating of the index lesion if focal therapy is being attempted. This uses high energy directional ultrasound (HIDU).
4. ExAblate Prostate: This is a transrectal MR guided device which is currently undergoing clinical trials. Calcifications 2 mm or greater in the ultrasound beam path and less than 5 mm from the rectal wall are a contra-indication.

Prostate calcifications are commonly found in elderly men, up to 50% by some estimates with higher incidence in men who have lower urinary tract symptoms. These are mostly made up of calcium apatite. They are mostly seen at the junction of transitional zone and peripheral zone with other locations being rare. Prostate calcifications can be seen as echogenic foci on ultrasound which may or may not shadow depending on their size. However, cross sectional information about the calcification is more beneficial especially while therapy planning. Computed tomography imaging is the current gold-standard for prostate calcification imaging. Current widely used MR techniques do not adequately image prostate calcifications. Calcifications are usually T1 and T2 dark but can be bright on both. T1 bright microcalcifications are noted frequently in the brain. Calcifications have also been shown to be bright on T2 weighted images (Fahr disease and chondrocalcinosis). The change in signal is thought to be related to closely associated water molecules in the microcalcification lattice. Gradient echo images cannot differentiate between calcifications and hemorrhage. There is definite need to develop and validate MR imaging techniques to visualize focal calcifications, especially for focal therapy planning and monitoring. It will obviate need for CT correlation, help in focal ablation modality selection and give true relative location of the calcification vis-à-vis visualized tumor without need for fusion. Imaging calcifications and evaluation of their effect on high energy ultrasound will help us define clinically significant calcifications. It is also the first step in development of techniques to mitigate effect of calcifications on therapeutic ultrasound.

3 promising MR techniques are available:

* A study by Zhu WZ et al., showed that both calcification and hemorrhage manifested low signal on susceptibility weighted images, but they presented opposite signal features on the corrected phase images. Significant difference was found in average phase shift between calcification and hemorrhage (t=74.69, p<0.05). These have been applied in the prostate before but size correlation has not been reported. An example of SWI imaging for calcification is provided.
* Zero-time echo (ZTE) and Ultra-short time echo (UTE) images have also been shown to image tissues with short T2 times like cortical bone. These can be used to study some stages of calcifications. To our knowledge, these have not been applied in the prostate before.
* Temperature uncertainty images can also be used to visualize calcifications in the prostate. This was observed in the currently undergoing clinical pivotal clinical trial of transurethral prostate ablation.

Comparison between these three MRI sequences, and the gold standard CT imaging of the pelvis will be performed to determine whether MRI can reliably identify and accurately measure the size of the prostate calcifications.

ELIGIBILITY:
Inclusion Criteria:

* Men 18 years and older
* prostate calcifications on CT obtained within the last 6 months

Exclusion Criteria:

* subjects with known prostate cancer
* subjects with any type of bioimplant, mechanical, electronic or magnetic means because such devices may be displaced or malfunction
* patients with cerebral aneurysm clips
* patient's with embedded shrapnel, metal workers, and machinists
* subjects who cannot adhere to the experimental protocols
* subjects who are not able to give consent
* subjects who exhibit claustrophobia or who exhibit severe vertigo when moved into the magnet.
* prisoners
* any other reason not included above, that would preclude the patient from obtaining an MRI

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Patient has to have a prostate.
Study Population: Men who are 18 years or older with prostatic calcifications on CT
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-09 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Size of calcifications | 1 day At time of CT or MRI
  Size of calcifications including volume on CT compared to each of the 3 MRI sequences

SECONDARY OUTCOMES:
Number of calcifications | 1 day At time of CT or MRI
  Number of prostate calcifications seen on CT and on MRI

CONTACTS AND LOCATIONS:
Overall Officials: Janesh Lakhoo, MD, Principal Investigator — Resident at Vanderbilt University Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhu WZ, Qi JP, Zhan CJ, Shu HG, Zhang L, Wang CY, Xia LM, Hu JW, Feng DY. Magnetic resonance susceptibility weighted imaging in detecting intracranial calcification and hemorrhage. Chin Med J (Engl). 2008 Oct 20;121(20):2021-5. PMID 19080268
- [Background] Tyler DJ, Robson MD, Henkelman RM, Young IR, Bydder GM. Magnetic resonance imaging with ultrashort TE (UTE) PULSE sequences: technical considerations. J Magn Reson Imaging. 2007 Feb;25(2):279-89. doi: 10.1002/jmri.20851. PMID 17260388
- [Background] Straub S, Laun FB, Emmerich J, Jobke B, Hauswald H, Katayama S, Herfarth K, Schlemmer HP, Ladd ME, Ziener CH, Bonekamp D, Rothke MC. Potential of quantitative susceptibility mapping for detection of prostatic calcifications. J Magn Reson Imaging. 2017 Mar;45(3):889-898. doi: 10.1002/jmri.25385. Epub 2016 Jul 15. PMID 27418017
- [Background] Bai Y, Wang MY, Han YH, Dou SW, Lin Q, Guo Y, Li W, Ding DG, Dai JP, Qin W, Shi DP, Tian J, Dai YM. Susceptibility weighted imaging: a new tool in the diagnosis of prostate cancer and detection of prostatic calcification. PLoS One. 2013;8(1):e53237. doi: 10.1371/journal.pone.0053237. Epub 2013 Jan 7. PMID 23308170
- [Background] Adams LC, Boker SM, Bender YY, Diederichs G, Fallenberg EM, Wagner M, Hamm B, Makowski MR. Diagnostic accuracy of susceptibility-weighted magnetic resonance imaging for the evaluation of pineal gland calcification. PLoS One. 2017 Mar 9;12(3):e0172764. doi: 10.1371/journal.pone.0172764. eCollection 2017. PMID 28278291
- [Background] Sundaram KM, Chang SS, Penson DF, Arora S. Therapeutic Ultrasound and Prostate Cancer. Semin Intervent Radiol. 2017 Jun;34(2):187-200. doi: 10.1055/s-0037-1602710. Epub 2017 Jun 1. PMID 28579687
- [Background] Hong CG, Yoon BI, Choe HS, Ha US, Sohn DW, Cho YH. The Prevalence and Characteristic Differences in Prostatic Calcification between Health Promotion Center and Urology Department Outpatients. Korean J Urol. 2012 May;53(5):330-4. doi: 10.4111/kju.2012.53.5.330. Epub 2012 May 18. PMID 22670192